CLINICAL TRIAL: NCT04076072
Title: High-speed Beveled Tip Versus Standard Tip Vitrectomy Probe: a Prospective Randomized Clinical Trial
Brief Title: Beveled-Tip Versus(vs) Standard-Tip Vitrectomy Probe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Shriji Patel, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 190728
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Results first posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-09

CONDITIONS: Vitrectomy
Keywords: vitrectomy

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial comparing the Ultravit High-Speed Beveled Probe with the current Alcon vitrector probe in a cohort of patients undergoing routine vitrectomy surgery.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization and data storage will occur in RedCap. Patients will be randomized the day of surgery by a masked study coordinator. The randomization numbers will be generated using the following procedure to ensure that treatment assignment is unbiased and concealed from patients and investigator staff. A patient randomization list will be produced by the IRT provider using a validated system that automates the random assignment of patient numbers to randomization numbers. These randomization numbers are linked to the different treatment arms. The randomization scheme for patients will be reviewed and approved by a member of the Randomization Group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Alcon Advanced Ultravit High-Speed Vitrectomy Probe (Active Comparator): On the day of surgery, patients will be randomized to the Ultravit High-Speed Beveled Probe or the current non-beveled Alcon Probe. All patients will undergo routine vitrectomy surgery as scheduled; patients will be unaware of the vitrector probe used. Time to completion of vitrectomy and time to completion of vitreous base shave will be recorded by study staff unaware of the vitrector probe used. All examination will be repeated as regularly scheduled postoperative visits by a reader unaware of which probe was used. Safety will be assessed at each visit by evaluation for any adverse events.
  Interventions: Device: Utravit High-Speed 10000 cpm Beveled Probe
- Alcon Non-Beveled Tip Vitrectomy Probe (Active Comparator): On the day of surgery, patients will be randomized to the Ultravit High-Speed Beveled Probe or the current non-beveled Alcon Probe. All patients will undergo routine vitrectomy surgery as scheduled; patients will be unaware of the vitrector probe used. Time to completion of vitrectomy and time to completion of vitreous base shave will be recorded by study staff unaware of the vitrector probe used. All examination will be repeated as regularly scheduled postoperative visits by a reader unaware of which probe was used. Safety will be assessed at each visit by evaluation for any adverse events.
  Interventions: Device: standard vitrector probe- Alcon (non-beveled) Ultravit 7500 cpm

INTERVENTIONS:
Device: Utravit High-Speed 10000 cpm Beveled Probe — This is a randomized controlled trial comparing the Ultravit High-Speed Beveled Probe with the current Alcon vitrector probe in a cohort of patients undergoing routine vitrectomy surgery.
  Arms: Alcon Advanced Ultravit High-Speed Vitrectomy Probe
Device: standard vitrector probe- Alcon (non-beveled) Ultravit 7500 cpm — This is a randomized controlled trial comparing the Ultravit High-Speed Beveled Probe with the current Alcon vitrector probe in a cohort of patients undergoing routine vitrectomy surgery.
  Arms: Alcon Non-Beveled Tip Vitrectomy Probe

SUMMARY:
The purpose of this study is to compare the efficiency of the new Utravit High-Speed 10000 cpm Beveled Probe to the current standard vitrector probe- Alcon (non-beveled) Ultravit 7500 cpm.

Study Design:

This is a randomized controlled trial comparing the efficiency of the Ultravit High-Speed Beveled Probe with the current Alcon vitrector probe in a cohort of patients undergoing routine vitrectomy surgery.

Hypothesis:

The Advanced Ultravit high-speed beveled probe will show non-inferiority to the standard, Alcon (non-beveled) Ultravit 7500 cpm with regards to time to completion of vitrectomy and surgical outcomes.

DETAILED DESCRIPTION:
High-speed beveled tip versus standard tip vitrectomy probe: a prospective randomized clinical trial

Background:

The Advanced Ultravit High-Speed Beveled Probe (Alcon) has a beveled-tip design that allows the cutting port to come closer to the retina compared to the previous vitrectr probe design. This allows the surgeon to maneuver in tight tissue planes and increases the functionality of the vitrector probe. This in combination with the increased cut rate of 10,000 independent cuts per minute reduces traction on the retina and increases efficiency of vitreous removal.

Purpose:

The purpose of this study is to compare the efficiency of the new Utravit High-Speed 10000 cpm Beveled Probe to the current standard vitrector probe- Alcon (non-beveled) Ultravit 7500 cpm.

Study Design:

This is a prospective, randomized controlled trial comparing the efficiency of the Advanced Ultravit High-Speed Beveled Probe with the current Alcon vitrector probe in a cohort of patients undergoing routine vitrectomy surgery.

Primary objectives:

-Intraoperative efficiency of vitrectomy surgery regarding time to completion of core vitrectomy and shave of vitreous base

Exploratory Objective:

-Intraoperative complications (e.g. iatrogenic retinal breaks, intraocular bleeding, retinal detachment)

Postoperative complications:

The study will not be sufficiently powered to assess safety. Surgeons will want to make sure there is no significant increase in complications with a different probe. However, any post operative complications would merely be an association, without any causality attributed.

Primary Endpoint:

A clinically significant difference in time to completion of core vitrectomy and shave of vitreous base between the two groups with 80% power at a 95% confidence interval.

A p-value of less than 0.05 will be deemed as statistically significant.

Sample Size Calculation Target: 40 participants (20 in each cohort) Assuming an average core vitrectomy time of 12 +/- 3 minutes, a sample size of at least 32 is needed to adequately assess for a clinically significant difference between the two groups with 80% power at a 95% confidence interval. A p-value of less than 0.05 will be deemed as statistically significant.

Procedures and Assessments:

All patients will undergo baseline testing in the study eye including:

* Best corrected Visual Acuity (BCVA)
* intraocular pressure (IOP)
* slit-lamp examination
* 360 degree indirect ophthalmoscopy

Enrollment Period:

9 months

Study Duration:

12 months

Methods:

On the day of surgery, patients will be randomized to the Ultravit High-Speed Beveled Probe or the current non-beveled Alcon Probe. All patients will undergo routine vitrectomy surgery as scheduled; patients will be masked to the vitrector probe used. Time to completion of vitrectomy and time to completion of vitreous base shave will be recorded by a masked timer.

All examination will be repeated as regularly scheduled postoperative visits by a masked reader.

Safety will be assessed at each visit by evaluation for any adverse events.

Randomization:

Randomization and data storage will occur in RedCap. Patients will be randomized the day of surgery. The randomization numbers will be generated using the following procedure to ensure that treatment assignment is unbiased and concealed from patients and investigator staff. A patient randomization list will be produced by the IRT provider using a validated system that automates the random assignment of patient numbers to randomization numbers. These randomization numbers are linked to the different treatment arms. The randomization scheme for patients will be reviewed and approved by a member of the Randomization Group.

Data collection measures:

* Unique Patient identifier
* Vision
* IOP
* Oculus sinister (Left Eye) /Ocular Dexter (Right Eye)
* Surgical Indication
* Time to completion of vitrectomy
* Time to completion of vitreous base shave
* Slit-lamp abnormalities
* Dilated Fundus Exam (DFE) abnormalities
* Post operation complications
* Data collection April 2019 to Dec 2019
* Data Analysis Jan 2020

Adverse Events:

Reporting of Adverse Events, Serious Adverse Events, and Unanticipated Problems Involving Risk to Participants or Others will be reported to the Institutional Review Board (IRB) pursuant to their policy as outlined under the VANDERBILT HUMAN RESEARCH PROTECTIONS PROGRAM Policy III.L.

Safety:

Risk Minimization:

The study will be conducted in accordance with the International Conference on Harmonization (ICH) along with the Good Clinical Practices (GCP) guidelines and all applicable local and U.S. federal regulatory requirements.

Prior to entry into the study or initiation of any study related procedures, the subject or legal representative must read, sign, and date the current institutional review board-approved version of the informed consent form. Fully informed consent or verbal consent must be obtained from the subject or legal representative in accordance with local legal requirements and IRB requirements.

Only potential subjects who meet the inclusion/exclusion criteria will be enrolled in to this protocol. The Principal Investigator will oversee all study procedures to ensure subject safety and protocol compliance.

Risk v. Benefits:

The prospective subject will be carefully screened to ensure inclusion/exclusion criteria are met.

There may be no direct benefit to the subjects ;however, the knowledge gained from this study may lead to improved methods of diagnosing, staging and managing Vitrectomy surgery in the future.

There will be no specific ethnic or age group targeted or excluded.

ELIGIBILITY:
Inclusion Criteria:

* The study population will be male and female patients 18 years old or older with the presence of pathology requiring routine vitreoretinal surgery (vitreous opacities, vitreous hemorrhage, vitreomacular traction, macular hole, epiretinal membrane) without previous history of vitreoretinal surgery. Ability to consent to procedure.

Exclusion Criteria:

* Previous incisional intraocular surgery other than uncomplicated cataract surgery with intraocular lens placement
* Inability to consent for procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shriji N Patel, MD, Principal Investigator — Vanderbilt Eye Institute
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 40 enrolled participants, 40 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | Alcon Advanced Ultravit High-Speed Vitrectomy Probe | Alcon Non-Beveled Tip Vitrectomy Probe
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 40 subjects including both male and female,18 years old or older, with the presence of pathology requiring vitreoretinal surgery (vitreous opacities, vitreous hemorrhage, vitreomacular traction, macular hole, epiretinal membrane) without previous history of vitreoretinal surgery.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcon Advanced Ultravit High-Speed Vitrectomy Probe | Alcon Non-Beveled Tip Vitrectomy Probe | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 10
  >=65 years | 13 | 17 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 8 | 11 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Pathology Requiring Vitreoretinal Surgery [Count of Participants; unit: Participants]
  Epiretinal Membrane | 2 | 3 | 5
  Vitreous Opacities or Hemorrhage | 10 | 13 | 23
  Vitreomacular Traction or Macular Hole | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Time to Completion of Core Vitrectomy and Shave of Vitreous Base
Description: Intraoperative efficiency of vitrectomy surgery regarding time to completion of core vitrectomy and shave of vitreous base
Time Frame: Time to completion of core vitrectomy and shave of vitreous base (12 ± 3 minutes )
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Alcon Advanced Ultravit High-Speed Vitrectomy Probe | Alcon Non-Beveled Tip Vitrectomy Probe
Number analyzed (Participants) | 20 | 20
minutes | 9.7 (2) | 10.4 (1.8)

2. Other Pre Specified Outcome: Number of Participants With Intraoperative Complications
Description: Participants in each study arm experiencing intraoperative complications (e.g. iatrogenic retinal breaks, intraocular bleeding, retinal detachment)
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Alcon Advanced Ultravit High-Speed Vitrectomy Probe | Alcon Non-Beveled Tip Vitrectomy Probe
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data is collected from study start to closure. Subjects are monitored for adverse effects through study completion, an average of 3 months.
Description: All AEs will be reported to PI and Alcon. Reporting of Adverse Events, Serious Adverse Events, and Unanticipated Problems Involving Risk to Participants or Others will be reported to the IRB pursuant to their policy as outlined under the VANDERBILT HUMAN RESEARCH PROTECTIONS PROGRAM Policy III.L.
Arm/Group | Alcon Advanced Ultravit High-Speed Vitrectomy Probe | Alcon Non-Beveled Tip Vitrectomy Probe
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT04076072/Prot_002.pdf
  • Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT04076072/SAP_003.pdf